CLINICAL TRIAL: NCT01423409
Title: Assessment of an Innovative Visual Analogue Scale of Pain (Pictorial VAS) Versus the Usual VAS (VAS) Among Deaf People
Brief Title: Multicenter Trial Assessing an Innovative VAS of Pain Among Deaf People
Acronym: EVA_SOURD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EVA SOURD study
Record Dates: First submitted 2011-07-22; First posted 2011-08-25 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-04

CONDITIONS: Deafness; Visual Analog Pain Scale
Keywords: visual analog pain scale; Deaf persons; clinical trial; multicentric
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pictorial VAS (Active Comparator): VAS with colours and 6 expressive faces
  Interventions: Device: pictorial VAS
- usual VAS (Sham Comparator): VAS
  Interventions: Device: usual VAS

INTERVENTIONS:
Device: pictorial VAS — Pictorial VAS includes elements which promote understanding of Deaf people: colours and 6 detailed expressive faces.
  Arms: pictorial VAS
Device: usual VAS — usual visual analog scale (VAS) of pain (line from 0: no pain to 10:worst pain)
  Arms: usual VAS

SUMMARY:
The purpose of this study is to assess an innovative Visual Analogue Scale of pain (pictorial VAS) versus the usual VAS (VAS) among Deaf People.

The assumption of this study is that pictorial VAS is more suited to Deaf people than usual VAS.

DETAILED DESCRIPTION:
Indeed French literature showed that 80% of Deaf people are illiterate. Moreover, lip-reading only allows to recognize one third of words.

Pictorial VAS includes elements which promote understanding of Deaf people: colours and 6 detailed expressive faces.

ELIGIBILITY:
Inclusion Criteria:

* people aged over 18 years old
* Deaf people
* affiliation to the french social security system or equivalent
* people who signed the consent form

Exclusion Criteria:

* hearing people
* people who became deaf
* pregnant or breastfeeding women
* people deprived of freedom
* people hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Innovative Visual Analogue Scale of Pain (Pictorial VAS) Versus the Usual VAS (VAS) Among Deaf People | one hour
  an innovative visual analogue scale of pain (pictorial vas) versus the usual vas (vas) among deaf people, at hospital, in terms of good understanding of pain

SECONDARY OUTCOMES:
Average scores of pain between the both groups: pictorial VAS versus usual VAS | one hour
  pain score
Analgesic treatment between the both groups : pictorial VAS versus usual VAS | one hour
  analgesic treatment
Pain score and analgesic treatment before and after French Sign Language (FSL) explanations | one hour
  pain score and analgesic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Mongourdin, PH, Principal Investigator — University Hospital, Grenoble
Locations (4):
- France (4):
  - University Hospital, Grenoble
  - University Hospital, Marseille
  - La Pitié-Salpêtrière, Paris
  - University Hospital, Strasbourg

REFERENCES:
- [Background] Dagron J. [Deafness and recourse to help, starting the dialog]. Soins. 2001 Dec;(661):37-9. No abstract available. French. PMID 12012932
- [Background] Dagron J .Les silencieux. Chroniques de vingt ans de médecine avec les Sourds. Editions : Presse Pluriel, Paris. 2008 ; 287 p.
- [Background] Delaporte Y. Chapitre 1 : Qui sont les Sourds, histoire d'un mot. In : Les Sourds, c'est comme ça. Editions de la Maison des sciences de l'homme, Paris 2002 ; 398 p.
- [Background] Gillot Dominique. Le Droit des Sourds. Juin 1998. (mis en ligne le date : http://www.sante.gouv.fr/).
- [Background] Loi n°2005-102 du 11 février 2005. Pour l'égalité des droits et des chances, la participation et la citoyenneté des personnes handicapées.
- [Background] Circulaire ministérielle n°DHOS/E1/DGS/SD1B/SD1C/SD4A/2006/90 du 2 mars 2006. La Charte de la personne hospitalisée.
- [Background] Circulaire N°99-84 du 11.02.1999. (Relative à la mise en place de protocole de prise en charge de la douleur).